CLINICAL TRIAL: NCT04983979
Title: A Multi Site, Placebo Controlled, Double Blind Randomised Clinical Trial Evaluating the Effectiveness of Sodium Zirconium Cyclosilicate Versus Placebo to Enable Safe Optimisation of RASi Therapy in Patients With Diabetic Kidney Disease.
Brief Title: The ORTIZ Study: Optimising RASi Therapy With SZC
Acronym: ORTIZ
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 136721
Record Dates: First submitted 2021-07-09; First posted 2021-07-30 (Actual); Results first posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: CKD; Diabetes Mellitus, Type 2; Hyperkalemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperkalemia | interventions — sodium zirconium cyclosilicate

STUDY DESIGN:
Intervention Model Description: A Multi site, placebo controlled, double blind randomised clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind randomised clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SZC (Experimental): 3 month treatment using Sodium zirconium cyclocilicate. Doses of 5 or 10g once daily will be used. The dose will be titrated according to potassium levels performed at clinic visits
  Interventions: Drug: Sodium Zirconium Cyclosilicate
- Placebo (Placebo Comparator): 3 month treatment using matched placebo. Doses of 5 or 10g once daily will be used. The dose will be titrated according to potassium levels performed at clinic visits
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium Zirconium Cyclosilicate — sachets of 5g or 10g given OD titrated to serum potassium
  Other Names: Lokelma
  Arms: SZC
Drug: Placebo — matched placebo given titrated according to potassium at a dose to 5 or 10g
  Arms: Placebo

SUMMARY:
The hypothesis is that 3 months' treatment with SZC versus placebo will enable RASi (Irbesartan) maximisation in a cohort of patients with diabetic kidney disease.

DETAILED DESCRIPTION:
Inhibiting the renin angiotensin (RAS) system has been the cornerstone of therapy for patients with proteinuric CKD for almost 2 decades, to slow the decline in renal function, delay the presence of dialysis and reduce cardiovascular events and death.

There is evidence in both the cardiac and renal literature that suggests that maximising the dose of RAS therapy leads to improved outcomes over smaller doses of RAS therapy.

Indeed, many of the studies on which we base our care use doses which are higher than what the majority of our patients are taking. Thus patients are being systemically undertreated by therapies which have been shown to have robust reno protection. With up to 80% of patients on RASi therapy are not on maximal RASi therapy , putting them at risk of a more rapid progression and poorer outcomes and increased healthcare costs.

An important reason for this is the presence or fear around hyperkalaemia. With reports of significantly increased rate of hyperkalaemia seen following increases in prescribing of RASi therapy. These concerns have lead NICE to recommend not starting patients on RASi therapy if their potassium is >5mmol/l, and KDOQI guidelines recommending consideration of stopping RASi therapy if serum potassium is >5.5mmol/l.

ACE inhibitors and angiotensin receptor blockers are thought to confer long term renal protection through reduction of proteinuria. The reduction in glomerular pressure is a major mechanism leading to a reduction in proteinuria, and hence renal protection, however as a consequence there will also an acute fall in eGFR. Therefore, when starting/up titrating ACEi/ARB it is expected that there will be an acute fall in eGFR, which is expected to be more than compensated for due to the subsequent long term renal protection. Indeed, current NICE guidelines do not suggest any alteration in management until the drop in eGFR is >25%.

There is a currently huge unmet need to optimise RASi therapy in those patients with hyperkalaemia.

There have been recent advances in novel therapeutics which can lower potassium in patients. One such agent is Sodium zirconium cyclosilicate (SZC).

SZC is a highly selective inorganic cation exchanger designed to entrap potassium in the intestine.

It has been shown to effective in lowering potassium in patients with heart failure, Diabetes, CKD and RASi therapy. With around a 1mmol/l fall in the serum potassium on those treated with SZC, compared to placebo.

In the 5-large clinical trials it appears efficacious, well tolerated and safe.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent
2. Adults ≥ 18years old
3. Type 2 Diabetes
4. CKD defined as eGFR 25-60ml/min
5. Albuminuria with uACR measured at >33.9.mg/mmol (300mg/g)
6. On a stable (>4 weeks) of sub-maximal RASi dose, defined as any ACE or ARB dose up to and including 50% of maximum dose with evidence of hyperkalaemia potassium level >5.0mmol/l OR not currently on RASi therapy due to documented issues of hyperkalaemia in the past necessitating RASi discontinuation

Exclusion Criteria:

1. Active malignancy
2. Patients who lack capacity to give informed consent
3. GI disturbance/chronic diarrhoea/stoma
4. Subjects with a life expectancy of less than 3 months.
5. Women who are pregnant, lactating, planning to become pregnant or unwilling to use effective methods of contraception during the study.
6. Presence of any condition which, in the opinion of the investigator, places the subject at undue risk or potentially jeopardizes the quality of the data to be generated including NYHA class III/IV.
7. History of acute eGFR fall with RASi therapy (>30% in eGFR on initiation of RASi therapy)
8. Known hypersensitivity or previous anaphylaxis to SZC or Irbesartan
9. Hypotension: BP <120/70mm/hg at screening despite no antihypertensive agent use
10. Uncontrolled Blood pressure: BP >170/110 at screening
11. Evidence of prolonged QT on ECG QTc(f)>550msec
12. History of QT prolongation associated with other medications that required discontinuation of that medication
13. Treatment with lithium, or dual blockade with ACEi and ARB or mineralocorticoid inhibitor
14. History of congenital long QT syndrome
15. Symptomatic or uncontrolled atrial fibrillation despite treatment, or asymptomatic sustained ventricular tachycardia. Subjects with atrial fibrillation controlled by medication are permitted
16. Current or recent (within 3 months) participation in a clinical trial involving an investigational medicinal product.
17. Current treatment with a potassium binder medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-06-17 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keiran McCafferty, Study Chair — Barts & The London NHS Trust
Locations (1):
- Kieran Mccafferty, London, Uk, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After patient enrolment, patients were checked for eligibility, then randomized to either Arm A or B if eligible.
  18 participants were consented for inclusion in ORTIZ. 7 participants failed screening as they did not meet the inclusion criteria. Two participants were not randomised despite being eligible. One participant was deemed to be unable to comply with the study schedule. The other was screened and found to be eligible 2 days prior to study termination so was not randomised.
Groups:
- Experimental: SZC: 3 month treatment using Sodium zirconium cyclocilicate. Doses of 5 or 10g once daily will be used. The dose will be titrated according to potassium levels performed at clinic visits
- Placebo Comparator: Placebo: 3 month treatment using matched placebo. Doses of 5 or 10g once daily will be used. The dose will be titrated according to potassium levels performed at clinic visits
Period: Overall Study
Arm/Group | Experimental: SZC | Placebo Comparator: Placebo
Started | 4 | 5
Completed | 4 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Total 9 participants
Groups:
- Sodium Zirconium Cyclosilicate (SZC): 3 month treatment using Sodium zirconium cyclocilicate. Doses of 5 or 10g once daily will be used. The dose will be titrated according to potassium levels performed at clinic visits
  Sodium Zirconium Cyclosilicate: sachets of 5g or 10g given OD titrated to serum potassium
- Total: Total of all reporting groups
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) | Placebo | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 1 | 3 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (9.5) | 58.0 (14.2) | 57.8 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 4 | 4 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 1 | 1 | 2
  Asian | 2 | 4 | 6
  Other | 1 | 0 | 1
Type of Medical Histpry [Number; unit: participants]
  Diabetes | 3 | 5 | 8
  Hypertension | 1 | 3 | 4
  Kidney disease | 1 | 4 | 5
  Other | 2 | 2 | 4
  Unknown | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients on Maximum Dose (300mg) Irbesartan Therapy at 12 Weeks Compared to Placebo
Description: Difference in proportion of patients on maximum dose (300mg) Irbesartan therapy at the end of 12 weeks compared to placebo. Proportion is calculated per arm as number of individuals on maximum dose Irbesatan therapy divided by the number of individuals in the study arm. The difference in proportion is calculated as experimental arm - placebo comparator arm.
Time Frame: Study end (week 12)
Population: Patients with diabetic kidney disease
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) | Placebo
Number analyzed (Participants) | 4 | 5
Participants
  Number of participants reaching maximum dose of irbesartan | 2 | 3
  Number of participants with no available data on irbesartan dose | 1 | 0
  Number of participants who did not reach maximum dose of irbesartan | 1 | 2
Statistical Analysis 1: Comparison: Sodium Zirconium Cyclosilicate (SZC) vs Placebo; Due to the small sample size only an estimate of the difference between study arms was generated. No hypothesis tests were completed; Test type: Other; Risk Difference (RD) = -0.10, 95% CI 2-sided [-0.752 to 0.552]

2. Secondary Outcome: Change in Potassium From Baseline at Each Time Point
Description: Difference in potassium from baseline at each study visit (weeks 1, 2, 4, 6, 8,12) calculated as a mean for each study visit.
Time Frame: At each study visit (weeks 1, 2, 4, 6, 8,12)
Population: Patients with diabetic kidney disease
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) | Placebo
Number analyzed (Participants) | 4 | 5
mmol/L
  Week 1 | -0.58 (0.53) | 0.06 (0.42)
  Week 2 | -0.03 (0.45) | 0.24 (0.54)
  Week 4 | 0.10 (0.23) | 0.08 (0.36)
  Week 6 | -0.10 (0.54) | 0.16 (0.23)
  Week 8 | 0.05 (0.52) | 0.16 (0.52)
  Week 12 | -0.50 (0.50) | 0.16 (0.48)
Statistical Analysis 1: Comparison: Sodium Zirconium Cyclosilicate (SZC) vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; Mean Difference (Final Values) = -0.66, 95% CI 2-sided [-1.97 to 0.65] — Only the mean difference for the study end (week 12) is presented here

3. Secondary Outcome: Change in the BP at the End of the Study From Baseline
Description: Difference in systolic and diastolic BP from baseline to end of study follow-up (week 12) calculated as a mean for each study visit.
Time Frame: Study end (week 12)
Population: Patients with diabetic kidney disease
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Sodium Zirconium Cyclocilicate: 3 month treatment using Sodium zirconium cyclocilicate. Doses of 5 or 10g once daily will be used. The dose will be titrated according to potassium levels performed at clinic visits
  Sodium Zirconium Cyclosilicate: sachets of 5g or 10g given OD titrated to serum potassium
Arm/Group | Sodium Zirconium Cyclocilicate | Placebo
Number analyzed (Participants) | 4 | 5
mmHg
  Systolic BP | -3.75 (26.80) | -28.90 (28.20)
  Diastolic BP | 1.38 (10.54) | -7.40 (12.75)
Statistical Analysis 1: Comparison: Sodium Zirconium Cyclocilicate vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; Mean Difference (Final Values) = 25.15, 95% CI 2-sided [-48.83 to 99.13] — Difference in change in systolic blood pressure between study arms
Statistical Analysis 2: Comparison: Sodium Zirconium Cyclocilicate vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; Mean Difference (Final Values) = 8.78, 95% CI 2-sided [-22.92 to 40.47] — Difference in change in diastolic blood pressure between study arms

4. Secondary Outcome: Proportion of Patients Who Have a Potassium of >6mmol/l, or >6.5mmol/l at Any Time During the Study
Description: Difference in proportion of patients who have a potassium of >6mmol/l,, or >6.5mmol/l at any time during the study. Proportion is calculated per arm as number of individuals with a maximum potassium across study follow-up of >6mmol/l or >6.5mmol/l divided by the number of individuals in the study arm. The difference in proportion is calculated as experimental arm - placebo comparator arm.
Time Frame: Cumulative across study follow-up, assessed at study end (week 12)
Population: Patients with diabetic kidney disease.
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) | Placebo
Number analyzed (Participants) | 4 | 5
Participants | 1 | 0
Statistical Analysis 1: Comparison: Sodium Zirconium Cyclosilicate (SZC) vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; Risk Difference (RD) = 0.25, 95% CI 2-sided [-0.174 to 0.674]

5. Secondary Outcome: Proportion of Patients Who Have a Potassium of <3.5mmol/l •
Description: Difference in proportion of patients who have a potassium of <3.5mmol/l at any time during the study. Proportion is calculated per arm as number of individuals with a minimum potassium of <3.5mmol/l across study follow-up divided by the number of individuals in the study arm. The difference in proportion is calculated as experimental arm - placebo comparator arm.
Time Frame: Cumulative across study follow-up, assessed at study end (week 12)
Population: Patients with diabetic kidney disease
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) | Placebo
Number analyzed (Participants) | 4 | 5
Participants | 0 | 0
Statistical Analysis 1: Comparison: Sodium Zirconium Cyclosilicate (SZC) vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; Risk Difference (RD) = 0.00, 95% CI 2-sided [0.00 to 0.00]

6. Secondary Outcome: Proportion of Patients Whose Glomerular Filtration Rate (GFR) Falls by >30% From the Previous Visit •
Description: Difference in proportion of patients with a sudden drop in GFR defined as >30% decreased between study visits. Proportion is calculated per arm as number of individuals experiencing a sudden drop of GFR divided by the number of individuals in the study arm. The difference in proportion is calculated as experimental arm - placebo comparator arm.
Time Frame: Cumulative. Calculated at each study visit. Assessed at study end (week 12).
Population: Patients with diabetic kidney disease
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) | Placebo
Number analyzed (Participants) | 4 | 5
Participants | 1 | 0
Statistical Analysis 1: Comparison: Sodium Zirconium Cyclosilicate (SZC) vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; Risk Difference (RD) = 0.25, 95% CI 2-sided [-0.174 to 0.674]

7. Secondary Outcome: Change in GFR at the End of Study From Baseline
Description: Difference in GFR from baseline to end of study follow-up (week 12) calculated as a mean for each study visit.
Time Frame: Study end (week 12)
Population: Patients with diabetic kidney disease
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) | Placebo
Number analyzed (Participants) | 4 | 5
mL/min/1.73m^2
  eGFR at Baseline | 41.00 (18.49) | 42.80 (12.58)
  eGFR at 12 weeks | 35.00 (16.19) | 40.80 (7.79)
  Difference from baseline | -6.0 (2.83) | -2.00 (7.28)
Statistical Analysis 1: Comparison: Sodium Zirconium Cyclosilicate (SZC) vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; Mean Difference (Final Values) = -4.0, 95% CI 2-sided [-19.5 to 11.4]

8. Secondary Outcome: Frequency of Adverse Events
Description: A count of the number of adverse events reported in each study arm
Time Frame: Study end (week 12)
Measure: Number; unit: adverse events across participants
Arm/Group | Sodium Zirconium Cyclocilicate | Placebo
Number analyzed (Participants) | 4 | 5
adverse events across participants | 6 | 6

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: AE: Any untoward medical occurrence in a participant to whom a medicinal product has been administered, including occurrences which are not necessarily caused by or related to that product.
  AEs that do not require reporting Specific biochemical and physiological parameters (potassium, BP, creatinine) will be expected to be altered as part of the predefined protocol and would not be expected to be reported as AEs: with the exception of those associated with an SAE or an AESI.
Arm/Group | Experimental: SZC | Placebo Comparator: Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/5
Other Adverse Events (participants affected / at risk) | 3/4 | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: SZC (N=4) | Placebo Comparator: Placebo (N=5)
Broken left humerus (Surgical and medical procedures) | 0 (0) | 1 (1) — Participant fell and broke their left humerus. This injury required a hospital admission for orthopaedic surgery. This SAE was deemed to be of moderate severity but was not deemed to be related to trial conduct, the IMP (SCZ/Placebo) or Irbesartan.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: SZC (N=4) | Placebo Comparator: Placebo (N=5)
Oedema (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Stomach Cramps (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Itchiness (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fluid overload (Endocrine disorders) | 0 (0) | 1 (1)
Weight gain (General disorders) | 0 (0) | 1 (1)
Worsening hypertension (Cardiac disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination due to unacceptably slow rate of recruitment. 9 participants were randomised. Extensive statistical analysis would not be proportionate, would not have meaningful statistical power, and would not be amendable to the drawing of inferences in respect of trial hypotheses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-07-05): https://cdn.clinicaltrials.gov/large-docs/79/NCT04983979/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-01): https://cdn.clinicaltrials.gov/large-docs/79/NCT04983979/SAP_001.pdf